CLINICAL TRIAL: NCT02033928
Title: Comprehensive Frailty Assessment
Status: Completed | Type: Observational
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Ashley Rosko, Principal Investigator, Ohio State University Comprehensive Cancer Center
Other Study IDs: OSU-13135
Record Dates: First submitted 2013-12-18; First posted 2014-01-13 (Estimated); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Myeloma, Multiple; Paraproteinemias; Hematologic Neoplasms
Keywords: Myeloma; MGUS (monoclonal gammopathy of undetermined significance); amyloidosis; stem cell transplant
MeSH Terms: conditions — Multiple Myeloma; Paraproteinemias; Hematologic Neoplasms; Neoplasms, Plasma Cell; Monoclonal Gammopathy of Undetermined Significance; Amyloidosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Arm I: Transplant patients
- Arm II: Plasma cell dyscrasia patients

SUMMARY:
The purpose of this research study is to describe a patients' fitness before and after treatment (whether that treatment be chemotherapy or a transplant). Fitness is a way of measuring a patient's current quality of health. With surveys, questionnaires and blood tests, we hope to create a tool that will give a good picture of patients' ability to tolerate treatment. In the future, we hope to devise the best treatment for a patient based on their "fitness".

ELIGIBILITY:
Inclusion Criteria:

* patients with a plasma cell dyscrasia AND/OR any patient receiving a stem cell transplant for a hematologic malignancy at The Ohio State University
* at least 18 years of age

Exclusion Criteria:

- Any medical or psychiatric condition that would make it difficult for the patient to comply with study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at The Ohio State University with a plamsa cell dyscrasia and/or any patient receiving a blood or marrow transplant at Ohio State will be considered for this study.
Sampling Method: Non-Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2014-04; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Change in Comprehensive Frailty Assessment | up to 14 months
  Responses to the Comprehensive Frailty Assessment will be assessed before and after treatment and changes will be evaluated. In transplant patients, this will be measured one year post transplant and in the non-transplant arm, this will be assessed after the second cycle of treatment.

SECONDARY OUTCOMES:
Time to progression | date of enrollment to date of documented clinical progression up to two years post-enrollment
  We will assess time to progression for multiple myeloma patients and the relationships of those outcomes to patients' functional, cognitive and psychosocial health.

OTHER OUTCOMES:
Overall survival | enrollment to date of death up to two years post-enrollment
  We will assess overall survival and the relationship of those measures to patients' functional, cognitive and psychosocial health.

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Rosko, MD, Principal Investigator — The Ohio State University Comprehensive Cancer Center
Locations (1):
- The Ohio State University Hospital East, Columbus, Ohio, United States

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu